CLINICAL TRIAL: NCT04253561
Title: A Phase Ib Study of Ipatasertib, an AKT Inhibitor, in Combination With Pertuzumab Plus Trastuzumab in Patients With PI3KCA-mutant, HER2-positive Locally Advanced or Metastatic Breast Cancer
Brief Title: Ipatasertib + Pertuzumab +Trastuzumab in Advanced HER2+ PI3KCA-mutant Breast Cancer Patients
Acronym: IPATHER
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-1507; 2019-001526-94 (EudraCT Number)
Record Dates: First submitted 2020-01-17; First posted 2020-02-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ipatasertib; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ipatasertib + Trastuzumab + Pertuzumab (Experimental): Ipatasertib will be given from Day 1 to Day 21 in every 28-day cycles. The starting dose is 400 mg orally (PO) QD and may be decreased to 300 mg QD and further to 200 mg QD (dose levels 1, - 1 and -2, respectively).
  Pertuzumab will be given IV every 21 days at the dose of 420 mg.
  Trastuzumab will be given SC every 21 days at the dose of 600mg. Intravenous (IV) Trastuzumab
  Interventions: Drug: Ipatasertib; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib will be administered orally once a day, beginning on Cycle 1, Day 1 through Day 21 of each 28-day cycle.
  Other Names: GDC-0068
Drug: Trastuzumab — 600 mg every 3 weeks
  Other Names: Herceptin
Drug: Pertuzumab — 420 mg every 3 weeks
  Other Names: Perjecta

SUMMARY:
This is an open label, single arm, multicenter, phase Ib study to evaluate the safety and clinical activity of the combination of ipatasertib, trastuzumab and pertuzumab in patients with unresectable locally advanced or metastatic HER2-positive breast cancer with tumors harboring PIK3CA mutations, candidates to receive maintenance HP after first line treatment for metastatic disease with a taxane plus HP

DETAILED DESCRIPTION:
The main objective of the study is to assess whether the combination of ipatasertib and HP (+/- ET) is tolerable, especially in terms of the incidence and severity of diarrhea. For this purpose, up to a total of 25 patients will be enrolled in a staggered manner and evaluated.

A 3-cohort, descending doses (400, 300, 200 mg) design will serve to establish the Maximun Toleraded Dose (MTD) and Recommended Phase 2 Dose (RP2D) of ipatasertib in combination with HP.

The study will initially include 6 patients that will receive ipatasertib plus HP at Dose Level 1.

If ≤1 DLTs are observed, this dose will be deemed safe, and the trial will enroll at least additional 19 patients to further assess safety and preliminary efficacy of the combination.

If ≥2 DLT occurs in the first 6 patients, a decision will be made of whether expand Dose Level 1 to 10 additional patients or to de-escalate ipatasertib to the next lower dose level. In the case of de-escalation, the same rules will apply for enrollment and expansion of Dose level -1. The minimum ipatasertib dose explored will be Dose level -2.

Dose reductions of pertuzumab and trastuzumab will not be allowed.

If all inclusion criteria and no exclusion criteria are met, patients will be enrolled in the trial and will start treatment with oral (PO) ipatasertib once a day (QD) D1-21 in 28-days cycles, together with pertuzumab 420 mg intravenous (IV) every 21 days (Q21d) and trastuzumab 600 mg subcutaneous (SC) Q21d.

Patients with hormone receptor positive (HR+) tumors (defined as ER and/or PgR expression in >1% of tumor cells) will also receive endocrine therapy either an Aromatase Inhibitor (AI), tamoxifen or fulvestrant +/- Luteinizing Hormone-Releasing Hormone (LHRH) analogues, according to Investigator's decision.

Patients will also start loperamide (2 mg twice a day [BID] or 4 mg QD) as prophylaxis for diarrhea in the first cycle

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent for all study procedures according to local regulatory requirements prior to beginning of specific protocol procedures.
2. Female (pre- or postmenopausal) or male patients.
3. Age ≥ 18 years.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
5. Confirmed HER2-positive invasive breast cancer by central determination defined by American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) clinical practice guidelines. (Wolff el al. Arch Pathol Lab Med-Vol 142, November 2018;).
6. Known hormone receptor status, as assessed locally, defined by ASCO/CAP clinical practice guidelines. ER/PR positivity is defined as the presence of ≥ 1% of tumor cells with nuclear staining (Hammond et al. JCO 2010).
7. Histologically confirmed, locally advanced or metastatic adenocarcinoma of the breast.

   1. Patients with unresectable locally advanced disease must have recurrent or progressive disease, which must not be amenable to resection with curative intent. Patients with available standard curative options are not eligible.
   2. For patients with bilateral breast cancer, HER2-positivity must be demonstrated in both locations or in a metastatic biopsy.
8. Patient must be a candidate to receive maintenance HP after first line treatment for metastatic disease with at least 4 cycles of taxane plus HP.
9. Prior taxane must have been discontinued for a reason other than progressive disease.
10. Patients may or may not have received neo/adjuvant therapy but must have a disease-free interval from completion of anti-HER2 therapy to metastatic diagnosis ≥6 months.
11. PIK3CA mutation identified and confirmed in tumor tissue or plasma ctDNA by central determination.
12. Start of treatment with ipatasertib plus HP no later than 9 weeks after last dose of taxane plus HP (i.e., maximum of 2 HP administrations with no taxane).
13. Willingness and ability to provide archived formalin fixed paraffin embedded (FFPE) tissue block.
14. Measurable or non-measurable (but evaluable) disease, as per RECIST 1.1 criteria.
15. No baseline diarrhea or diarrhea grade ≤1 within the last 28 days.
16. Adequate hematologic and organ function within 14 days before the first study treatment on Day 1 of Cycle 1, defined by the following:

    1. Neutrophils (ANC ≥1500/μL)
    2. Hemoglobin ≥9 g/dL (with no need for transfusions in the last 14 days).
    3. Platelet count ≥75,000/μL
    4. Serum albumin ≥3 g/dL
    5. Total bilirubin ≤1.5x the upper limit of normal (ULN), with the exception: patients with known Gilbert syndrome who have serum bilirubin ≤3x ULN.
    6. AST and ALT ≤2.5x ULN, with the following exception: patients with documented liver or bone metastases who may have AST and ALT ≤5x ULN.
    7. ALP ≤2x ULN, with the following exceptions:

       * Patients with known liver involvement who may have ALP ≤5x ULN.
       * Patients with known bone involvement who may have ALP ≤7x ULN.
    8. PTT (or aPTT) and INR ≤1.5x ULN (except for patients receiving anticoagulation therapy).

       * Patients receiving heparin treatment should have a PTT (or aPTT) between 1.5 and 2.5x ULN.
       * Patients receiving coumarin derivatives should have an INR between 2.0 and 3.0 assessed in two consecutive measurements 1 to 4 days apart.
    9. Serum creatinine <1.5x ULN or creatinine clearance ≥50 mL/min based on Cockcroft-Gault glomerular filtration rate estimation:

       (140 - age) x (weight in Kg) x 0.85 (if female)/72 x (serum creatinine in mg/dL)
    10. Fasting total serum glucose ≤150mg/dL and glycosylated hemoglobin (HbA1C) ≤7.5%
17. Life expectancy of at least 6 months.
18. Baseline left ventricular ejection fraction (LVEF) ≥50% measured by echocardiography (ECHO) or Multiple Gate Acquisition (MUGA) scan.
19. Negative β-HCG pregnancy test (serum) for premenopausal women of reproductive capacity (those who are biologically capable of having children) and for women less than 12 months after the menopause. All subjects who are biologically capable of having children must agree and commit to the use of a reliable method of birth control from 2 weeks before administration of the first dose of investigational product until 28 days after the last dose of investigational product.
20. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Exclusion Criteria:

1. Last dose of taxane plus HP given more than 9 weeks prior to C1D1.
2. Prior malignancy within 3 years prior to randomization, except curatively treated non-melanoma skin, carcinoma in situ of the cervix or Stage I uterine cancer.
3. Brain metastases that have not been treated previously, are progressive, or require any type of therapy (e.g., radiation, surgery, or steroids) to control symptoms within 30 days prior to the first study treatment dose.
4. Radiotherapy for metastatic sites of disease outside of the brain performed within 14 days prior to study enrollment and/or radiation of >30% of marrow-bearing bone.
5. Symptomatic hypercalcemia requiring use of bisphosphonate or RANKL inhibitors therapy within 21 days prior to the first study treatment. Patients who receive bisphosphonate therapy specifically to prevent skeletal events are eligible if they have been initiated prior to the treatment to study.
6. Cardiopulmonary dysfunction as defined by:

   1. Inadequately controlled angina or serious cardiac arrhythmia not controlled by adequate medication.
   2. Inadequate LVEF at baseline, as defined as LVEF <50% by either ECHO or MUGA scan.
   3. History of symptomatic congestive heart failure (CHF): Grade ≥3 per NCI CTCAE version 4.03 or Class ≥II New York Health Association (NYHA) criteria.
   4. History of a decrease in LVEF to <40% or symptomatic CHF with prior trastuzumab or HP treatment.
   5. History of myocardial infarction within 6 months prior to randomization.
   6. Current dyspnea at rest due to complications of advanced malignancy, or other disease requiring continuous oxygen therapy.
7. Congenital long QT syndrome or screening QT interval corrected using Fridericia's formula (QTcF) > 480 milliseconds.
8. Concurrent, serious, uncontrolled infections or current known infection with HIV (testing is not mandatory).
9. History of intolerance, including Grade 3-4 infusion reaction or hypersensitivity, to trastuzumab or pertuzumab.
10. Known hypersensitivity to any of the study drugs, including excipients.
11. Known clinically significant history of liver disease consistent with Child-Pugh Class B or C, including active viral or other hepatitis (e.g., positive for hepatitis B surface antigen [HBsAg] or hepatitis C virus [HCV] antibody at screening), current drug or alcohol abuse, or cirrhosis.

    * Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [HBcAg] antibody test) are eligible.
    * Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
12. History of Type I or Type II diabetes mellitus requiring insulin. Patients who are on stable dose of oral diabetes medication > 2 weeks prior to initiation of study treatment are eligible for enrollment.
13. Grade ≥2 uncontrolled or untreated hypercholesterolemia or hypertriglyceridemia.
14. History of or active inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis) or active bowel inflammation (e.g., diverticulitis).
15. Lung disease: pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, Aspergillosis, active tuberculosis, or history of opportunistic infections (Pneumocystis pneumonia or Cytomegalovirus pneumonia).
16. Need for chronic corticosteroid therapy of >10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids for a chronic disease.
17. Uncontrolled pleural effusion, pericardial effusion, or ascites. Patients with indwelling catheters (e.g., PleurX®) are allowed.
18. Treatment with strong CYP3A inhibitors or strong CYP3A inducers within 2 weeks or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study drug.
19. Prior treatment with an AKT inhibitor. Prior PI3K or mTOR inhibitors are allowed.
20. Current severe, uncontrolled systemic disease (e.g. clinically significant cardiovascular, pulmonary or metabolic disease; wound healing disorders; ulcers; bone fractures).
21. Unresolved, clinically significant toxicity from prior therapy, except for alopecia and Grade 1 peripheral neuropathy.
22. Major surgical procedure or significant traumatic injury within 28 days prior to enrollment.
23. Assessment by the investigator to be unable or unwilling to comply with the requirements of the protocol.
24. History of significant comorbidities that, in the judgment of the investigator, may interfere with the conduction of the study, the evaluation of response, or with informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
To define the Recommended Phase 2 Dose (RP2D) of ipatasertib when used in combination with HP (+/- ET) | From baseline to the end of cycle 1, up to 28 days
  The RP2D will be the dose level of ipatasertib at which no more than 1 subject of the study experiences a Dose Limiting Toxicity (DLT) defined by the protocol study.

SECONDARY OUTCOMES:
To evaluate the safety of the combination of ipatasertib with HP (+/- endocrine therapy [ET]). | Toxicities will be assessed during the whole treatment period (from baseline until lasts until 6 months after a patients' final treatment which is defined as the end of the Treatment Phase of the study).
  Number of patients with adverse events (AEs) and severe adverse events (SAEs) as per NCI CTCAE v4.03 of the combination of ipatasertib plus HP (+/- ET), with a special emphasis on the onset and severity of diarrhea.
To evaluate the tolerability of the combination of ipatasertib with HP (+/- endocrine therapy [ET]). | Toxicities will be assessed during the whole treatment period (from baseline until lasts until 6 months after a patients' final treatment which is defined as the end of the Treatment Phase of the study).
  Quantification of dose interruptions, reductions and dose intensity
Objective Response Rate (ORR) of the combination of ipatasertib with HP (+/- ET) as maintenance therapy after first line treatment for HER2-positive metastatic BC with a taxane plus HP. | From date of randomization to disease progression, death, unacceptable toxicity, consent withdrawal or study termination, whichever came first, assessed up to 20 months .
  Proportion of patients who have a complete response (CR) or partial response (PR), as determined by the investigator through use of RECIST v1.1.
Duration of Response (DoR) to the combination of ipatasertib with HP (+/- ET) as maintenance therapy after first line treatment for HER2-positive metastatic BC with a taxane plus HP. | From date of randomization to disease progression, death, unacceptable toxicity, consent withdrawal or study termination, whichever came first, assessed up to 20 months .
  Time from the first occurrence of a documented Objective Response (OR) to disease progression, according to RECIST v1.1, or death from any cause, whichever occurs first.
Clinical Benefit Rate (CBR) of the combination of ipatasertib with HP (+/- ET) as maintenance therapy after first line treatment for HER2-positive metastatic BC with a taxane plus HP. | From date of randomization to disease progression, death, unacceptable toxicity, consent withdrawal or study termination, whichever came first, assessed up to 20 months .
  Percentage of patients achieving confirmed CR, PR or stable disease (SD) for at least 24 weeks after the beginning of the study treatment by RECIST v1.1.
Progression-free survival (PFS) to the combination of ipatasertib with HP (+/- ET) as maintenance therapy after first line treatment for HER2-positive metastatic BC with a taxane plus HP. | From date of randomization to disease progression, death, unacceptable toxicity, consent withdrawal or study termination, whichever came first, assessed up to 20 months .
  Time from the commencement of study treatment (Day 1) to the occurrence of PD, as determined by the investigator via RECIST v1.1, or death from any cause, whichever occurs first.

OTHER OUTCOMES:
To identify putative predictive and prognostic molecular biomarkers (in plasma and/or tumoral tissue) that might be associated with the therapeutic activity of the combination of ipatasertib with HP (+/- ET). | From date of randomization to treatment discontinuation (up to 20 months)
  Correlation between tissue- and blood-based biomarkers (and clinical features (eg. Baseline features) with clinical activity of the combination of ipatasertib plus HP. Gene expression of PAM50 and 360 panel genes will be determined by the nCounter®Breast Cancer 360 Panel that includes 752 genes that cover established breast cancer diagnostic and research signatures as well as key pathways at the interface of the tumor, tumor microenvironment, and immune response. T
To identify molecular mechanisms of resistance to the study treatment by analyzing genomic DNA and gene expression in FFPE tumoral tissue before study treatment and after progression of disease (PD). | From date of randomization to treatment discontinuation (up to 20 months)
  DNA mutation analysis will be performed on tumor DNA samples to assess the predictive value of the most prevalent mutations in this breast cancer subtype. Next Generation Sequencing with Illumina will be used. DNA-seq of the most prevalent mutations including, but not limited to: TP53, ESR1, PIK3CA, AKT1, GATA3, PTEN and TBX3
  Gene expression of PAM50 and 360 panel genes will be also determined by the nCounter®Breast Cancer 360 Panel to identify mechanisms of resistance
To identify molecular mechanisms of resistance to the study treatment by analyzing circulating tumoral DNA (ctDNA) before study treatment and after progression of disease (PD). | From date of randomization to treatment discontinuation (up to 20 months)
  Genetic alterations will be evaluated in relevant genes in the PI3K/Akt pathway, including but not limited to PIK3CA and AKT1 as well as in TP53, ESR1, GATA3, ERBB2 and PTEN, amongst others. Identifying potential discordances in the PIK3CA/AKT1 status between tumor samples and ctDNA may help clarify the prognostic and predictive significance of PIK3CA/AKT1 mutations in patients with breast cancer treated with ipatasertib and PH.
To characterize the pharmacokinetics (PK) of ipatasertib and its metabolite G-037720 when administered in combination with HP (+/- ET): area under the plasma concentration time-curve (AUC) | At day 15 of Cycle 1 (each cycle is 28 days)
  All PK variables will be summarised using the following descriptive statistics:
  * Number of non-missing observations (N).
  * Arithmetic mean and its 90% CI, standard deviation, coefficient of variation (CV%) and standard error (SE).
  * Geometric mean (GM) and its 90% CI and GM CV%.
  * Minimum, median, maximum.
  Ipataserib plasma concentrations will be summarised for each scheduled sampling time point using descriptive statistics. Individual plasma concentration data versus time will be presented in a data listing and visualised as individual concentration-time plots.
To characterize the pharmacokinetics (PK) of ipatasertib and its metabolite G-037720 when administered in combination with HP (+/- ET): terminal half-life (t1/2) | At day 15 of Cycle 1 (each cycle is 28 days)
  All PK variables will be summarised using the following descriptive statistics:
  * Number of non-missing observations (N).
  * Arithmetic mean and its 90% CI, standard deviation, coefficient of variation (CV%) and standard error (SE).
  * Geometric mean (GM) and its 90% CI and GM CV%.
  * Minimum, median, maximum.
  Ipataserib plasma concentrations will be summarised for each scheduled sampling time point using descriptive statistics. Individual plasma concentration data versus time will be presented in a data listing and visualised as individual concentration-time plots.
To characterize the pharmacokinetics (PK) of ipatasertib and its metabolite G-037720 when administered in combination with HP (+/- ET): maximum observed plasma concentration (Cmax) | At day 15 of Cycle 1 (each cycle is 28 days)
  All PK variables will be summarised using the following descriptive statistics:
  * Number of non-missing observations (N).
  * Arithmetic mean and its 90% CI, standard deviation, coefficient of variation (CV%) and standard error (SE).
  * Geometric mean (GM) and its 90% CI and GM CV%.
  * Minimum, median, maximum.
  Ipataserib plasma concentrations will be summarised for each scheduled sampling time point using descriptive statistics. Individual plasma concentration data versus time will be presented in a data listing and visualised as individual concentration-time plots.
To characterize the pharmacokinetics (PK) of ipatasertib and its metabolite G-037720 when administered in combination with HP (+/- ET): minimal observed plasma concentration (Cmin) | At day 15 of Cycle 1 (each cycle is 28 days)
  All PK variables will be summarised using the following descriptive statistics:
  * Number of non-missing observations (N).
  * Arithmetic mean and its 90% CI, standard deviation, coefficient of variation (CV%) and standard error (SE).
  * Geometric mean (GM) and its 90% CI and GM CV%.
  * Minimum, median, maximum.
  Ipataserib plasma concentrations will be summarised for each scheduled sampling time point using descriptive statistics. Individual plasma concentration data versus time will be presented in a data listing and visualised as individual concentration-time plots.
To characterize the PK profile of pertuzumab and trastuzumab when administered in combination with ipatasertib (+/- ET): area under the plasma concentration time-curve (AUC) | At day 15 of Cycle 1 (each cycle is 28 days)
  Study of PK parameters of pertuzumab and trastuzumab when administered in combination with ipatasertib (+/- ET) and comparison to previously reported values.
  All PK variables will be summarised using the following descriptive statistics:
  * Number of non-missing observations (N).
  * Arithmetic mean and its 90% CI, standard deviation, coefficient of variation (CV%) and standard error (SE).
  * Geometric mean (GM) and its 90% CI and GM CV%.
  * Minimum, median, maximum.
  Trastuzumab and pertuzumab plasma concentrations will be summarised for each scheduled sampling time point using descriptive statistics. Individual plasma concentration data versus time will be presented in a data listing and visualised as individual concentration-time plots.
To characterize the PK profile of pertuzumab and trastuzumab when administered in combination with ipatasertib (+/- ET): terminal half-life (t1/2) | At day 15 of Cycle 1 (each cycle is 28 days)
  Study of PK parameters of pertuzumab and trastuzumab when administered in combination with ipatasertib (+/- ET) and comparison to previously reported values.
  All PK variables will be summarised using the following descriptive statistics:
  * Number of non-missing observations (N).
  * Arithmetic mean and its 90% CI, standard deviation, coefficient of variation (CV%) and standard error (SE).
  * Geometric mean (GM) and its 90% CI and GM CV%.
  * Minimum, median, maximum.
  Trastuzumab and pertuzumab plasma concentrations will be summarised for each scheduled sampling time point using descriptive statistics. Individual plasma concentration data versus time will be presented in a data listing and visualised as individual concentration-time plots.
To characterize the PK profile of pertuzumab and trastuzumab when administered in combination with ipatasertib (+/- ET): maximum observed plasma concentration (Cmax) | At day 15 of Cycle 1 (each cycle is 28 days)
  Study of PK parameters of pertuzumab and trastuzumab when administered in combination with ipatasertib (+/- ET) and comparison to previously reported values.
  All PK variables will be summarised using the following descriptive statistics:
  * Number of non-missing observations (N).
  * Arithmetic mean and its 90% CI, standard deviation, coefficient of variation (CV%) and standard error (SE).
  * Geometric mean (GM) and its 90% CI and GM CV%.
  * Minimum, median, maximum.
  Trastuzumab and pertuzumab plasma concentrations will be summarised for each scheduled sampling time point using descriptive statistics. Individual plasma concentration data versus time will be presented in a data listing and visualised as individual concentration-time plots.
To characterize the PK profile of pertuzumab and trastuzumab when administered in combination with ipatasertib (+/- ET): minimal observed plasma concentration (Cmin) | At day 15 of Cycle 1 (each cycle is 28 days)
  Study of PK parameters of pertuzumab and trastuzumab when administered in combination with ipatasertib (+/- ET) and comparison to previously reported values.
  All PK variables will be summarised using the following descriptive statistics:
  * Number of non-missing observations (N).
  * Arithmetic mean and its 90% CI, standard deviation, coefficient of variation (CV%) and standard error (SE).
  * Geometric mean (GM) and its 90% CI and GM CV%.
  * Minimum, median, maximum.
  Trastuzumab and pertuzumab plasma concentrations will be summarised for each scheduled sampling time point using descriptive statistics. Individual plasma concentration data versus time will be presented in a data listing and visualised as individual concentration-time plots.

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - ICO Badalona, Badalona, Barcelona
  - Comp. Hosp.Univ. Santiago (Chus), Santiago de Compostela, La Coruña
  - Hospital Universitario del Vall d' Hebron, Barcelona
  - H.Univ. Arnau de Vilanova de Lleida, Lleida
  - Centro Integral Oncológico Clara Campal (CIOCC), Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - MD Anderson, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Virgen de Macarena, Seville
  - Fundación Instituto Valenciano de Oncología, Valencia